CLINICAL TRIAL: NCT02882490
Title: Disruptive Behaviors in Children With Tourette Syndrome: the Role of Social Cognition and Efficacy of a Parent Behavioral Training Program
Brief Title: Parent Behavioral Training for Disruptive Behaviors in Tourette Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Spanish Association for Child and Adolescent Psychiatry (AEPNYA) (Unknown)
Responsible Party: Principal Investigator, Blanca Garcia-Delgar, M.D., Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AEPNYA 2014-2016
Record Dates: First submitted 2016-08-22; First posted 2016-08-29 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Tourette Syndrome; Behavioral Problem
Keywords: Tourette syndrome
MeSH Terms: conditions — Tourette Syndrome; Problem Behavior | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parent training (PT) (Experimental): The PT arm receives a 10-week therapist-guided behavioral group treatment. The treatment is based on existing literature for training parents in child behavior management skills (Barkley 1999). Parents attend weekly sessions, which last 90 minutes and are held at the Hospital Clinic of Barcelona. Parents are given homework assignments to complete between sessions.
  Interventions: Behavioral: Parent Training
- Supportive Therapy (ST) (Experimental): The ST arm receives a 10-week supportive group treatment. Parents are invited to discuss relevant problems that have occurred during the previous week. A therapist moderate the discussion but does not provide information about the behavioral techniques included in the PT group. Parents attend weekly sessions, which last 90 minutes and are held at the Hospital Clinic of Barcelona. Parents are given homework assignments to complete between sessions.
  Interventions: Other: Supportive Therapy

INTERVENTIONS:
Behavioral: Parent Training
  Arms: Parent training (PT)
Other: Supportive Therapy
  Arms: Supportive Therapy (ST)

SUMMARY:
This is a randomized controlled trial to assess the efficacy of a parent training program to control disruptive behaviors in children with Tourette Syndrome.

DETAILED DESCRIPTION:
Disruptive behaviors occur in 80% of children with Tourette Syndrome, and can be more disabling than the tics themselves.

The aim of this study is to assess the efficacy of a parent training program to control disruptive behaviors in children with Tourette Syndrome. In addition, social cognition will be examined in all the participants to analyze its relationship with the severity of disruptive behavior and the treatment response.

42 children with Tourette Syndrome and moderate disruptive behaviors will be randomly assigned to a 10-week Parent Training Program or a 10-week Supportive Therapy. Clinical response will be evaluated after the intervention period, and three and six months later.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill DSM-5 diagnostic criteria for Tourette's Disorder
* Moderate disruptive behaviors (Home Situations Questionnaire score >3)

Exclusion Criteria:

* Lifetime history of global learning disability, autism spectrum disorder, psychosis, bipolar disorder or organic brain disorder.
* Previous parent training with qualified therapist within the last 12 months prior to assessment
* Simultaneous individual treatment for disruptive behaviors.
* Initiation or adjustment of any psychotropic medication within the last 6 weeks prior to assessment

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2014-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Home Situations Questionnaire (HSQ) | Change from baseline to week 10; 3 months follow up; 6 months follow up
  Parent-rated scale with 16 items designed to assess behavioral non-compliance in regular home situations. Each item is rated on a 9-point Likert-type scale ranging from 1= "mild" to 9= "severe".

SECONDARY OUTCOMES:
Alabama Parenting Questionnaire | Change from baseline to week 10; 3 months follow up; 6 months follow up
  42-item clinical-administered questionnaire designed to measure the following dimensions of parenting style: 1- Positive involvement with children, 2- Supervision and monitoring, 3- Use of positive discipline technique, 4- Consistency in the use of such discipline and 5- Use of corporal punishment. Each item is scored on a 5-point, Likert-type scale from 1="never" to 5 = "always".
Parent Stress Index-Short Form | Change from baseline to week 10; 3 months follow up; 6 months follow up
  Parent-rated scale with 36-items questionnaire designed to measure stress in parent-child relationship.
The Gilles de la Tourette Syndrome-Quality of Life Scale (GTS-QOF) | Change from baseline to week 10; 3 months follow up; 6 months follow up
  Patient-reported scale with 27-items designed to measure health-related quality of life in children and adolescents with Tourette Syndrome.
Yale Global Tic Severity Scale (YGTSS) | Change from baseline to week 10; 3 months follow up; 6 months follow up
  Semi-structured interview to measure tic severity. After an initial inventory of current and lifetime motor and phonic tic types, current tic number, frequency, intensity, complexity and interference are rated on a 6-point scale. Maximum score is 100, resulting from three subscales: motor tic severity (maximum score 25), phonic tic severity (maximum score 25) and general impairment due to tics (maximum score 50).

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Morer, MD, Study Director — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sukhodolsky DG, Scahill L, Zhang H, Peterson BS, King RA, Lombroso PJ, Katsovich L, Findley D, Leckman JF. Disruptive behavior in children with Tourette's syndrome: association with ADHD comorbidity, tic severity, and functional impairment. J Am Acad Child Adolesc Psychiatry. 2003 Jan;42(1):98-105. doi: 10.1097/00004583-200301000-00016. PMID 12500082
- [Background] Barkley, R. A. (1999). Defiant teen: A Clinician's Manual for Assessment and Parent Training. New York: Guilford Press.